CLINICAL TRIAL: NCT02955992
Title: Guiding ICU Physicians' Communication and Behavior Towards Bereaved Relatives: a Randomized Controlled Trial (COSMIC - EOL)
Brief Title: Guiding ICU Physicians' Communication and Behavior Towards Bereaved Relatives
Acronym: COSMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AOM15014
Record Dates: First submitted 2016-11-03; First posted 2016-11-04 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Patients Died in Intensive Care Unit (ICU)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard of care (No Intervention)
- Intervention (Experimental): All caregivers will receive a leaflet about the importance of end of life (EOL) communication: key elements and recommendations regarding verbal and non-verbal communication.
  A "local champion" ("opinion leader") will be designated by each team in order to help implement the strategy. These physicians will help colleagues to connect external knowledge and requirements of the study to the local context.
  Development of a 3-step physician-driven support strategy starting after a decision to withhold or withdraw life-sustaining therapies is implemented:
  1. Preparation for the death : Prepare the relative for the patient's imminent death
  2. During the dying and death process: The physician enters the patient's room at least once to check on the relatives
  3. After the patient's death: the physician and the nurse meet the relative
  Interventions: Behavioral: Improving communication during the end-of-life process

INTERVENTIONS:
Behavioral: Improving communication during the end-of-life process
  Arms: Intervention

SUMMARY:
As ICU mortality is high, end-of-life is a subject of major concern for intensivists. With a mortality rate of 20%, end-of-life care has become a daily responsibility. Among those deaths, 60 to 80% follow a decision to withhold or withdraw treatment, situations where physicians, nurses and relatives must work together towards the most consensual decision. In this context, patients' relatives feel vulnerable and, in the months that follow the death, they are most likely to present symptoms that negatively affect their quality of life (anxiety, depression, PTSD, prolonged grief). Many studies have shown that communication with caregivers is one of the most highly valued aspects of care that impacts on family members' experience during the patient's stay and after the patient's death. Improving communication during the end-of-life process in the ICU context is a necessity that has been put forward in palliative care and family-centered care guidelines.

This study aims to improve both communication skills and behaviour by giving precise recommendations to physicians (3 step strategy) in their direct contact with patients' relatives. A 3-step physician-driven support strategy is used, that consists in 3 meetings with the relative - one before, one during and one after the patient's death. The underlying hypothesis is that this strategy will improve communication in the end-of-life setting and thus should reduce post-ICU burden for family members, specifically the development of prolonged grief 6 months after the death.

ELIGIBILITY:
Inclusion Criteria:

* Relatives of patients who died in the intensive care unit after a decision to withhold or withdraw treatment (adult ICUs only, ICU length of stay > 2 days).
* Consent to participate in the study
* Relative who was seen at least once by the physician before the patient's death

Exclusion Criteria:

* Relative that does not understand, read or speak French
* Relative who refuses to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
PG-13 : Prolonged Grief Disorder-13 that measures symptoms of prolonged grief | 6 months post patient's death

SECONDARY OUTCOMES:
CAESAR scale that measured quality of dying and death | 1 month post patient's death
Quality of dying and death (QODD-1) | 1 month post patient's ddeath
Miss-21 - Rapport subscale that describes communication with physician | 1 month post patient's death
Hospital Anxiety and Depression Scale (HADS) | 1, 3 and 6 months post patient's death
Impact of Event Scale-Revised (IES-R) that measures post-traumatic stress symptoms | 3 and 6 months post patient's death

OTHER OUTCOMES:
Questionnaire - lifestyle disruption | 6 months post patient's death
  Questionnaire developed by the Famiréa Group for relatives about lifestyle disruption
Checklist | 24 hours post patient's death
  Checklist for adherence of investigators to the intervention (intervention groups)

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Réanimation médicale Bicetre, Le Kremlin-Bicêtre, Val-de-marne
  - Anesthésie Réanimation Beaujon, Clichy
  - Réanimation polyvalente Sud Francilien, Évry
  - Réanimation Médicale hôpital Cochin, Paris
  - Réanimation médicale, Paris
  - Réanimation médicale Pitié Salpetriere, Paris
  - Réanimation chirurgicale HEGP, Paris
  - Réanimation médicale HEGP, Paris
  - Réanimation médico chirurgicale Tenon, Paris
  - Réanimation polyvalente René Dubos, Pontoise

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kentish-Barnes N, Chevret S, Valade S, Jaber S, Kerhuel L, Guisset O, Martin M, Mazaud A, Papazian L, Argaud L, Demoule A, Schnell D, Lebas E, Ethuin F, Hammad E, Merceron S, Audibert J, Blayau C, Delannoy PY, Lautrette A, Lesieur O, Renault A, Reuter D, Terzi N, Philippon-Jouve B, Fiancette M, Ramakers M, Rigaud JP, Souppart V, Asehnoune K, Champigneulle B, Goldgran-Toledano D, Dubost JL, Bollaert PE, Chouquer R, Pochard F, Cariou A, Azoulay E. A three-step support strategy for relatives of patients dying in the intensive care unit: a cluster randomised trial. Lancet. 2022 Feb 12;399(10325):656-664. doi: 10.1016/S0140-6736(21)02176-0. Epub 2022 Jan 19. PMID 35065008
- [Derived] Kentish-Barnes N, Chevret S, Azoulay E. Guiding intensive care physicians' communication and behavior towards bereaved relatives: study protocol for a cluster randomized controlled trial (COSMIC-EOL). Trials. 2018 Dec 22;19(1):698. doi: 10.1186/s13063-018-3084-7. PMID 30577862